CLINICAL TRIAL: NCT02838602
Title: Transnational Randomized Study Comparing Carbon Ions Therapy Versus Conventional Radiotherapy - Including Protontherapy - for the Treatment of Radioresistant Tumors
Brief Title: Randomized Carbon Ions vs Standard Radiotherapy for Radioresistant Tumors
Acronym: ETOILE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-760
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Malignant Tumors as Chordoma, Adenoid Cystic Carcinoma and Sarcoma
Keywords: carbon ions therapy; radiotherapy; radioresistant tumors; cancer; randomized trial
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Sarcoma; Neoplasms | interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon ions therapy (Experimental): Radical and exclusive carbon ions radiotherapy
  Interventions: Radiation: Carbon ions therapy
- Conventional radiotherapy (Active Comparator): Radical radiotherapy by Xrays and / or protons
  Interventions: Radiation: Advanced external radiotherapy by Xrays or protons

INTERVENTIONS:
Radiation: Carbon ions therapy — External radiotherapy by accelerated carbon nucleus in a specialized hadrontherapy center
  Arms: Carbon ions therapy
Radiation: Advanced external radiotherapy by Xrays or protons — Radiotherapy by any appropriate advance procedure of photontherapy (IMRT, Volumetric Modulated Arc Therapy (VMAT), Tomo, etc.) or when possible by protontherapy or even a combination of both types of radiotherapy
  Arms: Conventional radiotherapy

SUMMARY:
This is a transnational prospective randomized trial comparing definitive carbon ion therapy versus photon or combined photon and protontherapy as standard treatment for unresectable or macroscopically uncompleted resected radioresistant tumors. Eligible tumors are axial chordoma (except of base of skull), adenoid cystic carcinoma of head and neck (except of trachea) and sarcomas of any site (except chondrosarcoma of the skull base), non previously irradiated and without pre-planned surgery or chemotherapy after the clinical trial procedure. Randomization is balanced 1 for 1. Patients of the experimental arm are treated in carbon ions centers in Europe and patients of the standard arm are treated in France in their closest participating radiotherapy center. An accrual of 250 patients is needed and an absolute difference of 20% of relapse free survival at five years is awaited. The main endpoint is the progression free survival at five years. The trial is supported by the French program of clinical research and the national health insurance. Two associated studies are carried out: a radiobiological one looking for radioresistance markers in the sarcomas biopsies, and the second one is about medico economics.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* No severe comorbidity, life expectancy above 10 years
* Unresectable or inoperable or R2 resection of the tumor
* Eligible radioresistant tumor according to the limitative list as following:

  * adenoid cystic carcinoma of head and neck (larynx and trachea excluded)
  * soft tissue sarcoma
  * pleomorphic rhabdomyosarcoma only (alveolar and embryonal forms excluded)
  * retroperitoneal sarcoma under condition of technical feasibility (movement)
  * osteosarcoma of any grade and localisation (Ewing excluded)
  * chondrosarcoma (except of skull base) OMS grade >= 2
  * chordoma axial skeleton or pelvis (except of skull base)
  * angiosarcoma
* Absence of epidermal invasion (a hypodermic invasion is accepted with fixity of cutaneous plan but not true epidermal permeation)
* Larger volume to be irradiated (PTV) less than 25 cm
* ECOG Performance Status ≤ 2 or Karnovsky index ≥ 60
* no pregnancy of possibility of pregnancy during the treatment
* having an health insurance
* signature of a written informed consent
* validation of the randomization criteria: namely, a carbon ions therapy indication assessed by the medical team of a hadrontherapy center and able to by treated within two month from registration.

Exclusion Criteria:

* Complete macroscopic or microscopic surgical resection (R0 or R1)
* previous irradiation in the volume to be treated
* metastatic disease
* disease not candidate to a curative approach (example accelerated progressive diseaseresistant to nay medical treatment especially for sarcoma)
* any contra-indication to undergo a radiation therapy by Xray or particle therapy
* planned surgery or chemotherapy to take place after completion of radiotherapy (example : absence of enough space between an organ risk and the target volume (at least 5 mm) except the possibility of a spacer insertion)
* planned surgery or chemotherapy after radiotherapy
* Presence in the target volume of metallic material which cannot be removed (carbon fibres matreial authorized)
* history of concomittant (except in situ cervix carcinoma; or any cured basocellular cutaneous cancer tor any cured cancer with no sign of relapse during 5 years))
* impossible follow-up over 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-12-23 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to 5 years or loss of follow-up
  Starting point for PFS measurement is the randomization date

SECONDARY OUTCOMES:
Grades of the CTCAE-V4.02 classification | up to 5 years or loss of follow-up
  Tolerance
EQ-5D questionnaire | up to 5 years or loss of follow-up
  Quality of life
Local progression free survival | up to 5 years or loss of follow-up
  takes account of the local progression of the tumor in the planning target volume (PTV)
Metastases free survival | up to 5 years or loss of follow-up
  takes account of any site of relapse outside of the PTV
Overall survival | up to 5 years or loss of follow-up
  delay of death of any cause accounted starting from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Pascal POMMIER, MD, Principal Investigator — Centre Leon Berard
Locations (21):
- France (21):
  - CHU Amiens - Hôpital Sud, Amiens
  - Radiothérapie, CLCC François Baclesse, Caen
  - Radiothérapie, CRLCC Jean Perrin, Clermont-Ferrand
  - Radiothérapie, CRLCC GF Leclerc, Dijon
  - Radiothérapie, Hôpital A. Michallon, CHU de Grenoble, Grenoble
  - Radiothérapie, CRLCC Oscar Lambret, Lille
  - Radiothérapie, CRLCC Léon Bérard, Lyon
  - Radiothérapie, CRLCC Institut Paoli Calmettes, Marseille
  - Radiothérapie, Institut Régional du Cancer Montpellier, ICM Val d'Aurelle, Montpellier
  - Pôle de radiothérapie, Centre Antoine-Lacassagne, Nice
  - Radiothérapie, CHU Pitié-Salpétrière, Paris
  - Institut Curie, site Hôpital de Paris et site d'Orsay (Centre de protonthérapie), Paris
  - Radiothérapie, Hôpital de Haut Lévêque, CHU Bordeaux, Pessac
  - Radiothérapie, CRLCC Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Radiothérapie, CRLCC René Gauducheau, Saint-Herblain
  - Radiothérapie, Institut de Cancérologie de la Loire Lucien Neuwirtz, Saint-Priest-en-Jarez
  - Radiothérapie, CRLCC Paul Strauss, Strasbourg
  - Institut universitaire du cancer de Toulouse - Oncopole, Institut Claudius Regaud, Toulouse
  - Radiothérapie, Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
  - Radiothérapie, Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Balosso J, Febvey-Combes O, Iung A, Lozano H, Alloh AS, Cornu C, Herve M, Akkal Z, Lievre M, Plattner V, Valvo F, Bono C, Fiore MR, Vitolo V, Vischioni B, Patin S, Allemand H, Gueyffier F, Margier J, Guerre P, Chabaud S, Orecchia R, Pommier P. A randomized controlled phase III study comparing hadrontherapy with carbon ions versus conventional radiotherapy - including photon and proton therapy - for the treatment of radioresistant tumors: the ETOILE trial. BMC Cancer. 2022 May 23;22(1):575. doi: 10.1186/s12885-022-09564-7. PMID 35606739